CLINICAL TRIAL: NCT07398755
Title: A Prospective, Non-interventional, Single-Centre Study Assessing the Time Course of a Holistic Extended Periorbital Rejuvenation Procedure
Brief Title: Prospective, Non-interventional Study Assessing Periorbital Rejuvenation Procedure
Status: Active, not recruiting | Type: Observational
Sponsor: Yuvell (Other)
Collaborators: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: YUV-NIS-002
Record Dates: First submitted 2026-02-02; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Glabellar Lines; Midface Volume Deficiency; Periorbital Wrinkling
Keywords: Periorbital wrinkles; Facial wrinkles; Midface volume loss; Periorbital rejuvenation; Facial rejuvenation; Aesthetic dermatology
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Observational Cohort: Participants receiving routine clinical care/undergoing the rejuvenation procedure.
  Interventions: Drug: Letybo®; Device: Philart® Eye; Device: Saypha® Volume Plus Lidocaine

INTERVENTIONS:
Drug: Letybo® — Drug is used as part of routine clinical care. This observational study does not assign or modify treatment; it observes outcomes associated with drug use.
  Other Names: BoNT/A; botulinum toxin A; Letibotulinumtoxin A
Device: Philart® Eye — Device is used as part of routine clinical care. This observational study does not assign or modify treatment; it observes outcomes associated with device use.
  Other Names: polynucleotide
Device: Saypha® Volume Plus Lidocaine — Device is used as part of routine clinical care. This observational study does not assign or modify treatment; it observes outcomes associated with device use.
  Other Names: hyaluronic acid with lidocaine

SUMMARY:
The goal of this observation is to assess the time course of holistic extended periorbital rejuvenation using botulinum toxin A, cross-linked hyaluronic acid and polynucleotides corresponding to the application in routine practice in adults. It will also document the safety of treatment procedure and patient satisfaction.

The main questions it aims to answer are:

* How does a holistic extended periorbital rejuvenation procedure using botulinum toxin A, cross-linked hyaluronic acid filler, and polynucleotides change skin wrinkling around the eye area over time (particularly after 8 and 22 weeks)?
* How does the treatment affect the severity of dynamic glabellar lines at 8 and 22 weeks?
* Does the procedure improve midface volume deficiency after 8 and 22 weeks?
* How satisfied are participants with the overall rejuvenation treatment?

The investigator will observe the combination treatment of a drug Letybo® and medical devices PhilArt® Eye and Saypha® Volume Plus Lidocaine within their approved indications (non-interventional study, on-label use). The combination treatment aims to rejuvenate and improve the eye area holistically in patients coming routinely to the clinic.

Participants will:

* take PhilArt® Eye on Week 0 (Baseline), 3 and 6; Saypha® Volume Plus Lidocaine on Week 0 (Baseline); Letybo® on Week 6.
* visit the clinic on Week 0 (Baseline), 3, 6, 8 and 22 as per clinical practice for checkups and satisfaction assessment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older at time of treatment.
2. At least mild periorbital skin wrinkling, mild frown lines at maximum frown and mild.

   midface volume deficiency as assessed by the investigator
3. Subject has a stable medical condition with no uncontrolled systemic disease.
4. Willingness to participate in the routine follow-up after 8 weeks and 22 weeks and a signed informed consent form.
5. Subject already visiting the clinic for the specific treatment.

Exclusion Criteria:

1. Pregnancy and breast feeding.
2. Neuromuscular disease (e.g. myasthenia gravis, Eaton - Lambert syndrome).
3. Known impairment of blood coagulation.
4. Drooping eyelid.
5. Known allergy to botulinum toxin or human albumin (blood protein).
6. Presence of acute infection or inflammation at the proposed injection sites.
7. Botulinum toxin treatment in the glabella within the last 16 weeks.
8. HA- Filler treatment in the midface or periorbital area within the last 6 months.
9. Patients with a history of autoimmune disease or who are receiving immune therapy.
10. History of hypersensitivity to hyaluronic acid, lidocaine hydrochloride or other amidetype local anaesthetics.
11. History of fish product allergy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting the clinic for such a treatment as part of routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in skin wrinkling in periorbital area at Week 8 | Week 8
  Change in the percentage of skin wrinkling in the periorbital area from baseline to Week 8, as assessed using VISIA® skin analysis. Skin wrinkling is quantified as a percentage-based measurement derived from standardized VISIA imaging of the area around the eye. The outcome is expressed as the percent change relative to baseline, with higher percentages indicating an improvement, which equals a reduction in skin wrinkling.

SECONDARY OUTCOMES:
Change in skin wrinkling in the periorbital area at Week 22 | Week 22
  Change in the percentage of skin wrinkling in the periorbital area from baseline to Week 22, as assessed using VISIA® skin analysis. Skin wrinkling is quantified as a percentage-based measurement derived from standardized VISIA imaging of the area around the eye. The outcome is expressed as the percent change relative to baseline, with higher percentages indicating an improvement, which equals a reduction in skin wrinkling.
Change in severity of dynamic glabellar lines at Week 8 and Week 22 | Week 8, Week 22
  Change from baseline in everuty of glabellar lines at maximum frowning, measured at Week 8 and Week 22 using using the Facial Wrinkle Score (FWS).
  Severity of glabellar lines is quantified by comparing FWS scores at baseline and follow-up visits to assess severity grade during maximum frowning.
  The Facial Wrinkle Scale (FWS) is a validated photo-numeric scale ranging from 0 to 3, where higher scores indicate greater wrinkle severity.
Change from baseline in midface volume deficit severity, assessed at Week 8 and Week 22 by the investigator using the Midface Volume Deficit Severity Score (MVDSS) | Week 8, Week 22
  Change in investigator-assessed Midface Volume Deficit Severity Score (MVDSS) from baseline to Week 8.
  The MVDSS is used to evaluate the degree of midface volume deficiency based on clinical assessment. The outcome is expressed as the change in MVDSS score relative to baseline at each follow-up time point, with lower scores indicating a reduction in midface volume deficit severity.
  The Midface Volume Deficit Scale is a validated 5-point rating photo-numeric scale ranging from grade 0 to grade 4, where higher scores indicate greater very severe volume deficit.
Patient satisfaction with treatment assessed using a clinic-internal patient satisfaction questionnaire | Week 22
  Patient satisfaction with the treatment as assessed by participants using the clinic-internal questionnaire titled "Patient Satisfaction Questionnaire". The questionnaire consists of 5 questions evaluating the participant's overall satisfaction with the treatment outcome. Each item is rated on a numeric ordinal scale from 1 to 5, where lower scores indicate higher patient satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- YUVELL, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided